CLINICAL TRIAL: NCT04609748
Title: Comparative Analysis of the Effectiveness of the Use of Nimesulide and CBD Oil in Patients With Pain in the Preauricular Region Due to the Pain-dysfunctional Syndrome of the Temporomandibular Joint.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Dalewski Bartosz, Principal Investigator, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KB-0012/149/2020
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome; Temporomandibular Joint Pain
Keywords: temporomandibular joint; CBD oil; non steroid antyinflammatory drug; nimesulide
MeSH Terms: conditions — Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome | interventions — Cannabidiol; nimesulide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group that received nimesulide (Active Comparator)
  Interventions: Drug: Nimesulide
- The group that received CBD Oil (Experimental)
  Interventions: Drug: Cannabidiol Oil

INTERVENTIONS:
Drug: Cannabidiol Oil — Cannabidiol oil will be given twice a day, in a dose of 33,6mg, applied orally. The therapy will last 15 days.
  Arms: The group that received CBD Oil
Drug: Nimesulide — Nimessulid will be given twice a day - 2x100mg, applied orally. The therapy will last 15 days.
  Arms: The group that received nimesulide

SUMMARY:
During the study, the effectiveness of analgesic therapy with nimmsulide and cannabidiol oil will be compared.

Two study groups will be formed. The study will be conducted on patients reporting to the Dental Prosthetics Clinic of PUM in Szczecin. Patients aged 18-65 years with pain located in the area of the temporomandibular joint and the preauricular area, resulting from a dysfunction of the temporomandibular joint, will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (female and male) aged 18-65 years, able to swallow tablets
2. Patients with pain located in the temporomandibular and preauricular regions resulting from temporomandibular joint dysfunction
3. Patients with clinical diagnosis of Temporomandibular Joint Dysfunction

Exclusion Criteria:

1. patients with clinically diagnosed acute inflammation of the outer ear, middle ear, sinuses of the nose
2. patients allergic to nimesulide or cannabidiol oil
3. patients with contraindications to include therapy with nimesulide or cannabidiol oil such as:

   * gastric or duodenal ulcer disease,
   * severe blood clotting disorders,
   * severe liver dysfunction,
   * severe renal impairment,
   * severe heart failure, pregnancy,
   * breastfeeding,
   * concomitant intake of citrochrome blockers CYP3A4 or CYPP2D6 (warfarin, macrolides, calcium channel blockers, benzodiazepines, cyclosporine, sildenafil, SSRI, tricyclic antidepressants, opioids)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 15 days
  Measured on Visual Analogue Scale (VAS) scale. It consists of a line, approximately 100mm in length, at the left end of the scale "Score 0" which means "no pain", at the right end of the scale "Score 100mm" which means "worst imaginable pain"
Psychological conditions | 15 days
  Measured on The General Health Questionnaire-28 (GHQ-28)

CONTACTS AND LOCATIONS:
Locations (1):
- Chair and Depratment of Dental Prosthetics, Szczecin, Poland